CLINICAL TRIAL: NCT02853851
Title: Construction and Validation of a Stress Scale Specific to ICUs: Perceived Stressors in Intensive Care Units (PS-ICU)
Acronym: PS-ICU
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Laboratoire de psychologie université de franche Comté (Unknown); Unité de méthodologie et de qualité de vie en cancérologie CHU de besançon (Unknown); Hospital de Sabadell Department of Critical Care Spain (Unknown); Policlinico A. Gemelli Department of Critical Care Italy (Unknown); Centre hospitalier de l'Université de Montréal (CHUM) (Other); Alfred Hospital Intensive Care Unit Australia (Unknown)
Responsible Party: Sponsor
Other Study IDs: API/2014/56
Record Dates: First submitted 2016-07-20; First posted 2016-08-03 (Estimated); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Work Stress
Keywords: Stress factors,; intensive care units,; scale,; quality of care
MeSH Terms: conditions — Occupational Stress | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- France: 10 senior physicians, 10 interns, 10 experienced nurses (with more than one year of experience in the service) and 10 inexperienced nurses (with less than one year of experience in the service)
  Interventions: Other: interviews
- Italy: 10 senior physicians, 10 interns, 10 experienced nurses (with more than one year of experience in the service) and 10 inexperienced nurses (with less than one year of experience in the service)
  Interventions: Other: interviews
- spain: 10 senior physicians, 10 interns, 10 experienced nurses (with more than one year of experience in the service) and 10 inexperienced nurses (with less than one year of experience in the service)
  Interventions: Other: interviews
- montreal: 10 senior physicians, 10 interns, 10 experienced nurses (with more than one year of experience in the service) and 10 inexperienced nurses (with less than one year of experience in the service)
  Interventions: Other: interviews

INTERVENTIONS:
Other: interviews — Each subject will be asked to participate in an individual semidirective interview lasting about 40 minutes on the theme of the stress factors encountered in intensive care. All of the interviews will be audio-taped, transcribed and anonymized. The participants will also have to answer a socio-demographic questionnaire (sex, age, socio-professional category, speciality in intensive care, working hours, family situation, training, diplomas, length of time in the service).

SUMMARY:
This study aims to construct and validate an international professional perceived stress scale specific to intensive care units: the PS-ICU Scale (Perceived Stressors in Intensive Care Units).

DETAILED DESCRIPTION:
Intensive care units take charge of patients who present serious pathological states with an immediate vital risk in an emergency situation. Their treatment requires extensive coordination of human means and sometimes the use of complex procedures and technical means. Moreover, caregivers face the extreme situations of patients and their families coping with death, illness, pain and uncertainty (Weibel et al., 2003).

In this context, numerous stress factors that can have psychological consequences on the professionals and their effectiveness at work are inherent in intensive care (Donchin, 2002; Tummers et al., 2002).

In numerous studies, perceived stress proves to be more predictive of the subsequent health state of the individual than real stress (Consoli et al., 2001). More precisely, the authors have shown the influence of perceived stress on mental health (Ramirez et al., 1996b), psychical health (Chang et al., 2007), burnout (Bourbonnais et al., 1999), job dissatisfaction (Golbasi et al., 2008), absenteeism (Hackett & Bycio, 1996), turnover (Hayes et al., 2006) and more recently on the security of care (Endacott, 2012).

Identifying the factors of perceived stress is important in terms of mental health at work and the security of care. Studies on perceived stress have made it possible to elaborate stress scales specific to each profession (Borteyrou et al., 2013), with the aim of being as close as possible to the professionals' experience. However, to our knowledge, no stress scale for intensive care units has been published.

This study aims to construct and validate an international professional perceived stress scale specific to intensive care units: the PS-ICU Scale (Perceived Stressors in Intensive Care Units). Secondary objectives: To identify the factors of perceived stress having an impact on mental health, job satisfaction and the quality of care. To measure the impact of cultural and organizational dimensions on perceived stress in intensive care specific to each country. To measure the impact of socio-demographic variables on perceived stress. To measure the impact of coping abilities on perceived stress.

ELIGIBILITY:
Inclusion Criteria:

* In this step, we will include the services which:

  * Practise an activity of intensive care (whether this practice is medical or surgical, adult or paediatric).

The professionals of ICU who:

* volunteer to participate in the study (and with the consent of the head of the unit),
* Senior physicians, interns, and nurses who have been working in the service for more than three months.

Exclusion Criteria:

Administrative staff, nursing auxiliaries

* Senior physicians, interns, and nurses who have been working in the service for less than three months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The exploratory interviews will be conducted first in France. The French population will serve as the reference corpus, therefore the saturation threshold of the French reference corpus will determine the size of the corpus of the other countries (see the following section "analysis of the data").
  In each country, 10 senior physicians, 10 interns, 10 experienced nurses (with more than one year of experience in the service) and 10 inexperienced nurses (with less than one year of experience in the service) will be solicited for an exploratory interview.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
GENERATION OF ITEMS : Identifying the stress factors | up to 24 month
  In order to construct a first questionnaire based on all of the factors of perceived stress in intensive care, our research team will begin by identifying the stress factors. This identification will involve two main sources:

SECONDARY OUTCOMES:
GENERATION OF ITEMS: Selecting the items | up to 6 month
  All of the stress factors identified in the literature and in the exploratory interviews will then be grouped and organized according to the different dimensions of stress identified in health psychology
GENERATION OF ITEMS: Administering the PS-ICU questionnaire | up to 24 month
  The PS-ICU Questionnaire will be administered to a representative population (doctors and nurses in intensive care) in each of the countries involved. This population will allow us to do the analyses necessary for the reduction of the items, and to retain only the most reliable items. The administration of the questionnaire will also be used to evaluate several aspects: pertinence, comprehension, and redundancy of the items.
GENERATION OF ITEMS: Construction of the PS-ICU scale | up to 24 month
  Our research team will collect all of the quantitative data gathered in the framework of administering the PS-ICU questionnaire (France, Spain, Italia, Canada, Australia). It will be in charge of the statistical analysis and the interpretation of the results.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: Yes
eCRF